CLINICAL TRIAL: NCT06803329
Title: Qnnections: A Novel Suicide Prevention Intervention for Increasing Social Connection Among LGBTQ+ Veterans
Brief Title: Qnnections: Refinement and Pilot Trial of a Suicide Prevention Intervention to Increase Social Connection
Acronym: Qnnections
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: D5350-W; 1 IK2 RX005350-01A1 (Other: NIH)
Record Dates: First submitted 2025-01-27; First posted 2025-01-31 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Suicidal Thoughts and Behaviors; Social Isolation
Keywords: Suicide; Social isolation
MeSH Terms: conditions — Suicidal Ideation; Behavior; Social Isolation; Suicide

STUDY DESIGN:
Intervention Model Description: In Phase I (1.5 years), a pilot open trial (n = 10) will engage Veterans at elevated risk for suicide and gather acceptability data. Following refinement from Phase 1, Phase 2 (3.5 years) includes a pilot randomized feasibility and acceptability trial (n = 48), with participants randomized to Qnnections (10 group sessions, safety plan, referrals) or an Enhanced Usual Care condition that contains elements of standard VA suicide prevention (safety plan, referrals).
Who Masked: Outcomes Assessor
Masking Description: Assessors will be masked with regard to intervention condition to avoid bias, and participants will be instructed not to reveal their intervention condition. In Phase II, open-ended surveys will be used to collect qualitative data at post-treatment to allow for data collection without unmasking assessors.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Qnnections (Experimental): A novel group-based suicide prevention intervention that augments standard VA mental health services for LGBTQ+ Veterans with current suicidal thoughts or recent suicidal behavior. Veterans will also receive safety planning and referrals.
  Interventions: Behavioral: Qnnections
- Enhanced Usual Care (Active Comparator): The active control condition includes: 1) VA Safety Planning Intervention and 2) referrals to VA and non-VA services relevant to the individual.
  Interventions: Behavioral: Enhanced Usual Care

INTERVENTIONS:
Behavioral: Qnnections — A novel group-based suicide prevention intervention that augments standard VA mental health services for LGBTQ+ Veterans with current suicidal thoughts or recent suicidal behavior. Informed by the empirically-supported theoretical framework of the interpersonal theory of suicide and prior work tailoring interventions for minority stress, Qnnections is a structured 10-week group that uses a cognitive behavioral framework to target perceived burdensomeness and thwarted belongingness. Veterans will also receive safety planning and referrals.
  Arms: Qnnections
Behavioral: Enhanced Usual Care — The active control condition includes: 1) VA Safety Planning Intervention and 2) referrals to VA and non-VA services relevant to the individual. The safety plan will be conducted by Dr. Chang, a licensed psychologist. Therefore, EUC only differs from the Qnnections condition as it does not have the 10-session Qnnections intervention. EUC is intended to include elements of VA suicide prevention standard practice. The control condition is considered enhanced as all participants will receive these elements, whereas Veterans are not guaranteed to receive all of these services if not enrolled in this study.
  Arms: Enhanced Usual Care

SUMMARY:
Despite the high risk of suicide among LGBTQ+ Veterans, there is currently no suicide-focused intervention for this population. This study will refine and pilot Qnnections, a novel group-based suicide prevention intervention that aims to increase social connection and functioning in this population. The project will involve Veterans with lived experience in further refining Qnnections, and then will examine feasibility and acceptability of Qnnections and of study procedures in a pilot randomized clinical trial.

DETAILED DESCRIPTION:
Theoretical and empirical research consistently identifies perceived burdensomeness and thwarted belongingness as suicide-specific risk factors. This proposal refines and pilots Qnnections, a novel suicide prevention intervention which aims to increase social connection and functioning through improving belongingness and reducing burdensomeness. Phase I (1.5 years) focuses on intervention refinement of Qnnections with a Veteran Advisory Board (n = 8) and expert mentors. In its current form, Qnnections is a 10-week group-based intervention intended to augment Veterans Affairs (VA) suicide prevention efforts, using a cognitive behavioral framework to target social disconnection. After refinement by mentors and Veterans with lived experience, a pilot open trial (n = 10) will engage Veterans and gather acceptability data. Following refinement from Phase 1, Phase 2 (3.5 years) includes a pilot randomized feasibility and acceptability trial (n = 48), with participants randomized to Qnnections (10 group sessions, safety plan, referrals) or an Enhanced Usual Care condition that contains elements of standard VA suicide prevention (safety plan, referrals). Veteran participants in both phases will complete quantitative assessments at baseline, mid-treatment, post-treatment, and ten-week follow-up. Qualitative data collection will occur at post-treatment. The focus is feasibility and acceptability of Qnnections and of study procedures.

ELIGIBILITY:
Inclusion Criteria:

* Veterans who report past-month active suicidal ideation (C-SSRS [Columbia-Suicide Severity Rating Scale]

  -- or past-3-month suicidal behavior;
* LGBTQ+ or other minoritized gender or sexual identity;
* Have a mental health point-of-contact (e.g., Suicide Prevention Coordinator, Mental Health Treatment Coordinator);
* Willing to complete or update safety plan.

Exclusion Criteria:

* cannot provide informed consent;
* imminent psychiatric hospitalization;
* current or planned participation in residential/intensive outpatient program that would interfere study participation;
* in a conservatorship; and
* has participated in any previous parts of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2030-09-30 (Estimated); Study Completion 2030-09-30 (Estimated)

PRIMARY OUTCOMES:
Acceptability of Intervention Measure (AIM) | 10-20 weeks
  Weiner BJ, Lewis CC, Stanick C, et al. Psychometric assessment of three newly developed implementation outcome measures. Implementation Sci. 2017;12(1):108.
  4 items on a 5-point Likert scale from 1-5, with higher scores indicating greater acceptability, appropriateness, or feasibility. This scale has demonstrated promising psychometric properties for the monitoring and evaluation of an intervention's feasibility and acceptability. These measures are available in the public domain.
Intervention Appropriateness Measure (IAM) | 10-20 weeks
  Weiner BJ, Lewis CC, Stanick C, et al. Psychometric assessment of three newly developed implementation outcome measures. Implementation Sci. 2017;12(1):108.
  4 items on a 5-point Likert scale from 1-5, with higher scores indicating greater acceptability, appropriateness, or feasibility. This scale has demonstrated promising psychometric properties for the monitoring and evaluation of an intervention's feasibility and acceptability. These measures are available in the public domain.
Feasibility of Intervention Measure (FIM) | 10-20 weeks
  Weiner BJ, Lewis CC, Stanick C, et al. Psychometric assessment of three newly developed implementation outcome measures. Implementation Sci. 2017;12(1):108.
  4 items on a 5-point Likert scale from 1-5, with higher scores indicating greater acceptability, appropriateness, or feasibility. This scale has demonstrated promising psychometric properties for the monitoring and evaluation of an intervention's feasibility and acceptability. These measures are available in the public domain.

OTHER OUTCOMES:
Interpersonal Needs Questionnaire (INQ) | 10-20 weeks
  Van Orden KA, Cukrowicz KC, Witte TK, et al. Thwarted belongingness and perceived burdensomeness: Construct validity and psychometric properties of the Interpersonal Needs Questionnaire. Psychological Assessment. 2012;24(1):197-215.
  15-item self-report measure that has separate scales for perceived burdensomeness and thwarted belongingness, two social disconnection constructs from the well-established Interpersonal Theory of Suicide. The INQ has demonstrated both reliability and validity, and it has been used across diverse samples of sexual minority adults (Feinstein et al., 2022).
Beck Suicidal Ideation Scale (BSSI) | 10-20 weeks
  Beck AT, Steer, R. A. Manual for the Beck Scale for Suicide Ideation. Vol 63.; 1991.19-item interviewer-administered assessment of suicidal ideation severity. The total score may range from 0 to 38, with higher scores indicating greater suicidal ideation. The BSSI has demonstrated strong reliability and validity.
Patient-Reported Outcomes Measurement Information System (PROMIS) - Ability to Participate in Social Roles & Satisfaction with Ability to Participate in Social Roles | 10-20 weeks
  Hahn EA, DeWalt DA, Bode RK, et al. New English and Spanish social health measures will facilitate evaluating health determinants. Health Psychology. 2014;33(5):490-499.
  Two four-item questionnaires from the widely used PROMIS: Ability to Participate in Social Roles and Activities (PROMIS-APS) and the Satisfaction with Ability to Participate in Social Roles and Activities (PROMIS-SPS). Both subscales have scores ranging from 4-20, with higher scores indicating greater social functioning. Studies suggest these measures are responsive to change in diverse clinical populations.

CONTACTS AND LOCATIONS:
Overall Officials: Cindy Chang, PsyD, Principal Investigator — VA San Diego Healthcare System, San Diego, CA
Locations (1):
- VA San Diego Healthcare System, San Diego, CA, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No